CLINICAL TRIAL: NCT01307735
Title: Prospective Assessment of the Clinical Utility of Cardiovascular Magnetic Resonance in Patients With Suspected Acute Myocarditis - A Pilot Study for Establishing an International Registry
Brief Title: International Myocarditis Registry
Acronym: mmr
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Libin Cardiovascular Institute of Alberta (Other)
Responsible Party: Matthias Friedrich, Libin Cardiovascular Institute of Alberta
Other Study IDs: 232447
Record Dates: First submitted 2011-03-02; First posted 2011-03-03 (Estimated); Last update posted 2011-03-03 (Estimated); Status verified 2011-02

CONDITIONS: Myocarditis
Keywords: myocarditis; edema; hyperemia; fibrosis; necrosis; cardiovascular magnetic resonance imaging
MeSH Terms: conditions — Myocarditis; Edema; Hyperemia; Fibrosis; Necrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biopsy samples with viral or bacterial DNA
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Myocarditis negative on CMR: Patients with suspected myocarditis referred for CMR and not fulfilling at least 2 of the 3 CMR criteria (Lake Louise Criteria)for myocarditis.Lake Louise Criteria are edema, hyperaemia, and necrosis/fibrosis.
- Myocarditis positive on CMR: Patients with suspected myocarditis referred for CMR and fulfilling at least 2 of the 3 CMR criteria (Lake Louise Criteria)for myocarditis.Lake Louise Criteria are edema, hyperaemia, and necrosis/fibrosis.

SUMMARY:
Myocarditis is an inflammatory heart disease primarily of viral origin that can lead to heart failure and death. Despite an unfavorable long-term outcome and mortality rate as high as 50%, classification, diagnosis, and treatment of myocarditis remains controversial. The gold standard for clinical diagnosis is direct sampling of the heart muscle, which often misses the infected area and thus reliability of the test is questionable. While the cause and clinical presentation of myocarditis are often unclear, inflammation of the heart muscle can be clearly imaged by Cardiovascular Magnetic Resonance Imaging (CMR).

Due to recent international consensus on CMR protocol for myocarditis and the unique ability of CMR to visualize cardiac structure, function, and characterize tissue, CMR has become the primary tool for clinical assessment. This study aims to test the accuracy of CMR in the diagnosis of myocarditis and to validate whether CMR acquired in an early stage of myocarditis can provide incremental prognostic information. In order to effectively gather relevant clinical data, an online, multi-centre international registry will be established across twenty different medical institutions.

Hypotheses:

1. CMR accurately detects active myocardial inflammation in patients with myocarditis
2. CMR acquired in an early clinical stage of myocarditis provides incremental prognostic information superior to standard clinical diagnostic tools.

DETAILED DESCRIPTION:
Study Rationale Because of its unique combination of morphological and functional imaging with tissue characterization, cardiovascular magnetic resonance (CMR) has become the non-invasive diagnostic tool of choice for assessing myocarditis. Recently, standard diagnostic CMR criteria for myocarditis have been proposed ("Lake Louise Criteria"), based on signal intensity patterns in T2-weighted images and T1-weighted images before and after contrast administration 3.

There is however a lack of prognostic data using these criteria. Furthermore, the clinical utility of these criteria in a real-life scenario is not well understood.

The aim of the study is to evaluate the diagnostic CMR criteria for the prediction of functional outcome and quality of life in patients with myocarditis.

Background: Myocarditis Myocardial inflammation, most often caused by myocardial involvement in systemic viral illness, although typically of benign outcome, may result in persisting myocardial damage. Clinical outcomes include heart failure and death. Chronic myocarditis can progress to dilated cardiomyopathy which result in dilation and decompensation of one or both ventricles resulting in heart failure, with the need for cardiac transplantation.

Diagnostic approach to myocarditis The diagnosis of myocarditis is generally considered after exclusion of other causes of acute heart disease and established by a combination of history, physical examination with non-invasive or invasive tests.

History and clinical examination have to precede further diagnostic testing although the initial onset of myocarditis often is insidious, symptoms are non-specific, and clinical signs absent.

ECG findings, such as ST changes, AV block or arrhythmias may be associated with myocarditis, although their sensitivity is limited.

Serological biomarkers of myocardial injury such as creatine kinase and troponin may be increased; however, the prevalence of an increased troponin T in biopsy-proven myocarditis is limited, likely due to the lack of extensive necrosis in many cases.

Endomyocardial biopsy (EMB) usually is considered the gold standard in definitively diagnosing myocarditis. In 1986, a group of pathologists defined EMB criteria for the diagnosis of myocarditis, known as "The Dallas Classification System". This classification suggested that a minimum of three, but recommended that five separate biopsy specimens had to be taken for accurate pathological analysis. A major limitation of this technique is that it is invasive, with a mortality rate of 0.4% and certain contraindications9. Myocardial injury caused by viral infection could also have a focal distribution, which EMB may not be able to detect. Only 10 to 25% of patients with clinically suspected myocarditis have confirmed diagnosis by EMB11. High interobserver variability in the interpretation of EMB, and with the associated sampling errors, the clinical value of this technique is questioned.

Indium-111(111In)-antimyosin antibody (AMA) scintigraphy uses specific antibodies targeted at damaged myocytes, and thus, is able to detect in vivo necrosis. A major drawback of this technique, however, is that it cannot differentiate between different etiologies of myocardial necrosis. It is also not suitable to detect inflammation in the absence of cell death.

Prognostic value of diagnostic markers There is a paucity of data on the prognostic value of the various diagnostic tools. LV dysfunction is considered the most important indicator for worse outcome in myocarditis. In recent studies, however, LV dysfunction was infrequently observed3; therefore, this marker may not be helpful in most clinical scenarios, especially in less severe cases with persisting symptoms despite preserved cardiac function.

Background: Cardiovascular Magnetic Resonance (CMR) Hallmark features of acute myocarditis are interstitial lymphocytic infiltration with edema and hyperemia, and myocardial necrosis3. Interestingly, these can be readily identified by CMR in a non-invasive approach, using a combination of non-contrast and Gadolinium-enhanced techniques.

CMR offers several advantages, as opposed to other diagnostic modalities. It does not use radiation or harmful contrast agents, the field of view is not limited and tissue characterization can be combined with functional assessment of the ventricles in the same session.

The first clinical study using contrast-enhanced magnetic resonance imaging in patients with acute myocarditis showed that CMR is a suitable tool to detect myocardial inflammation and showed a spread of tissue changes from focal to diffuse myocardial involvement.

Based on previous pilot data, the same group further introduced T2-weighted CMR imaging in acute myocarditis as a specific marker for myocardial edema.

Areas of Gd accumulation in CMR images acquired late after contrast administration ("Late enhancement") reflect irreversible injury and were reported in about 60% of reported myocarditis cases.

The diagnostic sensitivity of a comprehensive CMR protocol is 67%, with a specificity of 91% and a diagnostic accuracy of 78%, which exceeds that of other diagnostic approaches. As sub-clinical myocarditis is also an immune response phenomenon, it is speculated that CMR parameters used for diagnosing acute myocarditis will also be relevant for imaging sub-clinical myocarditis. CMR is increasingly accepted as the emerging standard diagnostic test for myocarditis.

Prognostic CMR data in myocarditis Follow-up data on CMR in myocarditis are still scarce. In a pilot study, Wagner et al. studied the evolution of the relative enhancement in the early course of the disease and after months in patients with myocarditis compared with 26 healthy patients. They demonstrated that myocardial contrast enhancement decreases to normal values in many patients within a follow-up of 30 months. In 2/19 patients, left ventricular function did not recover. Interestingly, contrast enhancement on day 28 was predictive of the ejection fraction and of clinical outcome after 30 months.

More recently, Zagrosek et al. provided CMR follow-up data on 36 patients 18±10 months after myocarditis. They demonstrated that in the acute phase, T2 ratio and relative enhancement was elevated in most of the patients (86% and 80% respectively) and significantly decreased at follow-up, this was associated with improvement both in clinical and left ventricular function parameters. Late enhancement was present in 22 patients (63%) and persisted in 21/22 patients. The acute phase T2 ratio correlated significantly with the change in end-diastolic volume.

The predictive value of each of the CMR markers for inflammation (hyperemia, edema) and necrosis/fibrosis, however, is not known, especially when compared to LV function at presentation.

Study Objectives

1. The primary objective will be to compare CMR criteria for myocarditis at presentation with LV volumetric and functional outcome markers as acquired in a follow-up CMR study in patients with diagnostic CMR criteria for myocarditis and in a control group.
2. Secondary objective will be to compare compare CMR criteria for myocarditis at presentation with quality of life at 12 months after presentation in the same groups.

Study Variables

1. CMR Criteria for Myocarditis ("Lake Louise Criteria")

   Evidence for myocardial inflammation will be present if at least 2 of 3 CMR criteria are positive. These include:
   * Early Gd enhancement ratio equal to or greater than 4.0;
   * regional or global T2 signal intensity ratio equal to or greater than 2.0;
   * at least one focus of late enhancement.
2. LV function

   * Ejection fraction,
   * LVEDV,
   * LVESV,
   * LVEDVI,
   * LVESVI,
   * Stroke volume,
   * Cardiac index,
   * End-systolic wall stress
3. Quality of life will be quantified by a standardized questionnaire

Study Design Patients referred for a CMR study at the Stephenson Cardiovascular MR Centre for suspected myocarditis will be screened. Patients with CMR-derived evidence for myocarditis (i.e. at least two positive Lake Louise Criteria in at least one CMR scan during the clinically acute phase of the disease) will be considered "myocarditis-positive".

As a control group, patients referred for suspected myocarditis but not fulfilling the diagnostic CMR criteria for myocarditis and with normal systolic LV function. Both groups will receive the same standard protocol as per the Consensus Group recommendations.

Follow-up will be performed between 4 and 8 weeks after the initial episode and at 1 year. Data will include CMR results and quality of life assessment as quantified by a standardized questionnaire.

Subjects

Recruitment

1. Inpatients identified by study nurses in collaboration with supervising cardiologists
2. Outpatients in Cardiology clinics Imaging protocol

All CMR imaging will be performed on a 1.5T MRI system (Avanto®, Siemens Medical Solutions, Erlangen, Germany), with the use of a 32-channel cardiac phased array coil for functional and late enhancement images and the body coil for T2-weighted images and early Gd enhancement images. The protocol will be performed as follows:

* Left ventricular function Steady-state free precession (SSFP) gradient echo sequence Six rotational long axis views, with each slice thickness of 10mm, and zero spacing in between slices will be performed to cover the entire left ventricle.
* T2 weighted imaging Short TI inversion recovery (STIR) spin echo sequence Three short axis slices will be obtained at basal, mid, and apical regions. Each slice will be 15mm thick.

At this point, gadolinium-DTPA will be injected intravenously.

* Early enhancement imaging T1-weighted turbo spin echo sequence Three short axis slices will be obtained at basal, mid, and apical regions before and immediately after (over 4 minutes) administration of 0.1ml/kgBW Gd-DTPA. Each slice is 10mm thick, and the acquisition is T1-weighted and free-breathing. If image quality is insufficient in short axis views, axial slices will be acquired.
* Late enhancement imaging Inversion-recovery prepared gradient echo sequences with individual determination of inversion time according to maximal suppression of myocardial signal, a stack of short axis views and a set of rotational long axis views will be acquired 10 minutes after Gd-DTPA infusion. All of the left ventricle will be covered in short-axis slices.

ELIGIBILITY:
Inclusion Criteria:

1. At least 2 positive CMR criteria for myocarditis as acquired by a CMR study within less than 10 days of the onset of symptoms suggestive of myocarditis (fever, symptoms of systemic viral disease)
2. Evidence for cardiac involvement (elevated troponin, arrhythmia and/or ECG changes)

Exclusion Criteria:

1. Contraindication to CMR, such as implanted metal object, reaction to gadolinium, or severe claustrophobia
2. Acute or severe renal insufficiency (rapid increase of creatinine or creatinine clearance of ≤ 30ml/min)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred for a CMR study at the Stephenson Cardiovascular MR Centre for suspected myocarditis will be screened. Patients with CMR-derived evidence for myocarditis (i.e. at least two positive Lake Louise Criteria in at least one CMR scan during the clinically acute phase of the disease) will be considered "myocarditis-positive".
  As a control group, patients referred for suspected myocarditis but not fulfilling the diagnostic CMR criteria for myocarditis and with normal systolic LV function. Both groups will receive the same standard protocol as per the Consensus Group recommendations.
Sampling Method: Probability Sample
Enrollment: 78 (Estimated)
Dates: Start 2010-01; Primary Completion 2011-04 (Estimated); Study Completion 2011-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Matthias G Friedrich, MD, Principal Investigator — University of Calgary
Locations (1):
- Stephenson CMR Centre, Calgary, Alberta, Canada